CLINICAL TRIAL: NCT06152185
Title: Mindfulness App Training for Cardiovascular Health
Acronym: MATCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Thomas Kamarck, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY22090002; R34HL163245 (NIH)
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular Diseases; Mindfulness
Keywords: Mindfulness; Cardiovascular Disease; Stress
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the Mindfulness intervention (n = 63) or Enhanced Usual Care (n = 42) using a 3:2 randomization sequence.
Who Masked: Outcomes Assessor
Masking Description: The research associates who interact with participants following randomization will be blind to condition. The study coordinator and investigators will not be blind to condition; they will be responsible for interacting with participants during the intervention but will not be involved in post-randomization data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness Training (Experimental): Mindfulness intervention involving 28 audio-guided lessons plus daily brief practice prompts. Lessons train meditation techniques for 3 mindfulness skills: concentration, sensory clarity, and equanimity. Practice prompts delivered 3x daily build on the skills trained in each lesson.
  Interventions: Behavioral: Mindfulness Training
- Enhanced Usual Care (EUC) (Active Comparator): Participants in the EUC condition will have no study requirements during the 4-week intervention period, but they will receive a list of stress management resources upon randomization (websites, books, health tracking apps, and mental health services) with no additional intervention support.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Mindfulness Training — The mindfulness intervention includes 28 daily 20-minute audio lessons plus brief daily practice prompts. The first 14 lessons train techniques for developing foundational mindfulness skills through didactics and guided practice; the second 14 lessons review these techniques through guided practice. Based on the Unified Mindfulness system, lessons train 3 mindfulness skills: concentration, sensory clarity, and equanimity. Concentration, a state of stable attention, enables participants to monitor present-moment physical and emotional body experiences. Sensory clarity, the monitoring of momentary experiences, involves detecting subtle sensations and discriminating between different experiences. Equanimity, an attitude of acceptance toward momentary experiences, is trained through 3 strategies: (a) body relaxation, (b) mental welcoming, and (c) a gentle tone of voice. Practice prompts delivered 3 times daily encourage participants to practice brief moments of mindful awareness.
  Arms: Mindfulness Training
Behavioral: Enhanced Usual Care — Participants in the EUC condition will have no study requirements during the 4-week intervention period, but they will receive a list of stress management resources upon randomization (websites, books, health tracking apps, and mental health services) with no additional intervention support.
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
This study will investigate the feasibility and effects of a smartphone-based mindfulness training program vs. usual care in a sample of stressed midlife and older adults at risk for cardiovascular disease. 105 participants will be randomly assigned to complete a four-week mindfulness training intervention, which involves 28 audio-guided lessons and practice prompts delivered 3x daily, or to continue with their regular routines. Data will be collected at baseline, post-intervention, and three-month follow-up. The study will involve seven laboratory visits, which will include assessments and training on daily life monitoring and intervention procedures. Data assessing subjective and physiological stress reactivity in daily life will be collected for 3 days at pre-intervention, post-intervention, and 3-month follow-up. Passive sensor data will be continuously collected from participants' smartphones and wearable devices to develop models that predict daily life stress. Data will be used to evaluate feasibility of the intervention and assessments in a sample at risk for cardiovascular disease and to test effects of mindfulness training on subjective and physiological stress reactivity.

DETAILED DESCRIPTION:
This study is aimed at assessing the feasibility and effects of a smartphone-based mindfulness training program vs. usual care. The objective is to determine the program's effectiveness in reducing stress levels and cardiovascular responses to stress in the daily lives of participants, with a specific focus on individuals at risk of cardiovascular disease. Participants will be aged 45 or above and have risk factors for cardiovascular disease.

Participants will be randomly assigned to either receive a smartphone-based mindfulness training program or continue their regular daily routines. The study consists of seven laboratory visits that include assessments and training for completing at-home study activities and using monitoring devices. These devices will track activity levels, heart rate, and various stress indicators during the study at three separate weeklong periods.

A mobile blood pressure device will take hourly blood pressure readings during three monitoring days at pre-intervention, post-intervention, and three-month follow-up. On these days, participants will complete brief surveys on their smartphones at each reading and at the beginning and end of each day about their mood, behaviors, and social interactions. Participants will also wear Fitbit activity monitors and a sensor application will be installed on participants' smartphones to continuously collect data on movement, heart rate, location, screen status, and other parameters. Together, this data will be used to gain insights into daily stress indicators.

Participants assigned to the mindfulness training group will engage in daily 20-minute audio recordings and practice assignments at home over a one-month period. They will also be asked to answer questions about their daily stressors and the effectiveness of the training program, both at the beginning and end of each day. The study team will periodically contact them by phone to address any questions or concerns during this month. Participants assigned to the usual care control group will receive resources for stress management but will not participate in a structured intervention or be required to respond to specific questions over the one-month period.

After the intervention period, all participants will complete a second week of daily life monitoring, and a third week of monitoring three months later. They will also complete a laboratory cardiovascular reactivity task at pre-intervention and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 years or older
* Fluent in English and proficient in reading English
* Living in the Pittsburgh area for the next 5 months and available for study visits and activities during this period
* High perceived stress (greater than or equal to 14 on the 10-item Perceived Stress Scale)
* Diagnosed with hypertension by medical provider and, if medicated, blood pressure below 150/100, or if unmedicated, clinic blood pressure reading greater than or equal to 125/75 and less than 150/100
* Moderate-to-high cardiovascular disease risk, as indicated by hypertension and at least 1 of the following:

  * Diagnosed with diabetes by medical provider
  * Diagnosed with high cholesterol by medical provider
  * Current smoker by self-report (smoking or vaping every day or nearly every day)
  * Body Mass Index ≥30
* Android or iOS smartphone that meets study requirements
* Participant otherwise able to meet study requirements

Exclusion Criteria:

* Clinical or symptomatic atherosclerotic disease, including ischemic heart disease, heart failure, angina, stroke, or atrial fibrillation
* Two or more "night shift" episodes in the past month
* Pregnancy
* Typical alcohol consumption ≥15 drinks per week
* Marijuana or hashish use >9 of the past 30 days
* Use of other controlled substances (e.g., cocaine, crack, heroin, meth, ecstasy) in the past 30 days
* Current moderate-to-severe depressive symptoms (score ≥15 on PHQ-9)
* Suicidal ideation (PHQ-9 item 9 score >0)
* Positive PTSD screen (traumatic event(s) endorsed and total score ≥3 on Primary Care PTSD screen for DSM-5)
* Positive Bipolar Disorder screen (≥7 yes responses to item 1, yes to item 2, and moderate or serious on item 3 of Mood Disorder Questionnaire)
* Positive screen for psychosis (≥1 on Two-Item Screen for Early Psychosis)
* Regular systematic mind-body practice (e.g., yoga or meditation >2 times/week)
* Current participation in another clinical trial or in a study that uses smartphone software

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Task Strain from pre-intervention to post-intervention | Change in Task Strain assessed for 3 days at pre-intervention and post-intervention (an average of 5 weeks)
  Task strain assessed as the proportion of hourly observations during each ambulatory monitoring period that are assigned ratings above the sample median on a 3-item Task Demand scale and below the sample median on a 2-item Decision Latitude scale, with higher scores indicating higher task strain
Change in Task Strain from pre-intervention to 3-month follow-up | Change in Task Strain assessed for 3 days at pre-intervention and three-month follow-up (an average of 18 weeks)
  Task strain assessed as the proportion of hourly observations during each ambulatory monitoring period that are assigned ratings above the sample median on a 3-item Task Demand scale and below the sample median on a 2-item Decision Latitude scale, with higher scores indicating higher task strain
Change In Systolic Blood Pressure Response to Momentary Psychosocial Stress from pre-intervention to post-intervention | Change in Systolic Blood Pressure Response to Momentary Psychosocial Stress assessed for 3 days at pre-intervention and post-intervention (an average of 5 weeks)
  Ambulatory systolic blood pressure response in relation to hourly measures of momentary strain (high task demand and low decision latitude)
Change In Systolic Blood Pressure Response to Momentary Psychosocial Stress from pre-intervention to 3-month follow-up | Change in Systolic Blood Pressure Response to Momentary Psychosocial Stress assessed for 3 days at pre-intervention and three-month follow-up (an average of 18 weeks)
  Ambulatory systolic blood pressure response in relation to hourly measures of momentary strain (high task demand and low decision latitude)
Change in Social Conflict from pre-intervention to post-intervention | Change in Social Conflict assessed for 3 days at pre-intervention and post-intervention (an average of 5 weeks)
  Social conflict assessed hourly using a 3-item scale, with average scores ranging from 0-10 and higher scores indicating greater social conflict, and a 1-item exploratory measure, with scores ranging from 0-10 and higher scores indicating greater social conflict
Change in Social Conflict from pre-intervention to 3-month follow-up | Change in Social Conflict assessed for 3 days at pre-intervention and three-month follow-up (an average of 18 weeks)
  Social conflict assessed hourly using a 3-item scale, with average scores ranging from 0-10 and higher scores indicating greater social conflict, and a 1-item exploratory measure, with scores ranging from 0-10 and higher scores indicating greater social conflict
Change in Systolic Blood Pressure Response to Social Conflict from pre-intervention to post-intervention | Change in Systolic Blood Pressure Response to Social Conflict assessed for 3 days at pre-intervention and post-intervention (an average of 5 weeks)
  Ambulatory systolic blood pressure response in relation to hourly measures of social conflict
Change in Systolic Blood Pressure Response to Social Conflict from pre-intervention to 3-month follow-up | Change in Systolic Blood Pressure Response to Social Conflict assessed for 3 days at pre-intervention and three-month follow-up (an average of 18 weeks)
  Ambulatory systolic blood pressure response in relation to hourly measures of social conflict
Feasibility of recruitment | Assessed at enrollment
  Recruitment benchmark: >7 participants will be enrolled each month on average
Feasibility of retention | Assessed across the entire 5-month study period
  Retention benchmark: ≥73% retention from initial enrollment through follow-up
Feasibility of adherence | Assessed across the entire 5-month study period
  Adherence benchmark: average completion of ≥85% of intervention lessons and ≥75% of ambulatory assessments
Acceptability: Treatment Expectancies | Treatment Expectancies assessed among participants randomized to the mindfulness condition at pre-intervention, post-intervention (average of 5 weeks), and 3-month follow-up (average of 19 weeks)
  Acceptability of mindfulness intervention with benchmark of ≥75% of participants giving positive ratings of treatment expectancies (>3 on a 6-item Credibility/Expectancy Questionnaire, with higher scores indicating greater positive treatment expectancy)
Feasibility of safe implementation: Side Effects | Adverse effects assessed among participants randomized to the mindfulness condition at pre-intervention, post-intervention (average of 6 weeks), and 3-month follow-up (average of 20 weeks)
  Feasibility of safe implementation, with a benchmark of <10% of mindfulness participants endorsing occasional or moderately distressing side effects, assessed via the Adverse Effects Survey, a 15-item self-report survey on the frequency of unwanted side effects that may be associated with the experience of meditation
Acceptability: Study Burden | Study Burden assessed at post-intervention and 3-month follow-up
  Study burden benchmark of ≥80% of participants giving ratings of 2.5 (less than burdensome) or below on average on a 5-item measure of study load

SECONDARY OUTCOMES:
Change in Clinic Blood Pressure from pre-intervention to post-intervention | Change in clinic blood pressure assessed with 2 pre-intervention assessments and 2 post-intervention assessments (average of 6 weeks)
  Average of clinic blood pressure (systolic and diastolic) readings at two assessments for each time point (pre-intervention, post-intervention)
Change in Clinic Blood Pressure from pre-intervention to 3-month follow-up | Change in clinic blood pressure assessed with 2 pre-intervention assessments and 2 3-month follow-up assessments (average of 19 weeks)
  Average of clinic blood pressure (systolic and diastolic) readings at two assessments for each time point (pre-intervention, 3-month follow-up)
Change in Mean Ambulatory Blood Pressure from pre-intervention to post-intervention | Change in Mean Ambulatory Blood Pressure assessed for 3 days at pre-intervention and post-intervention (an average of 5 weeks)
  Average of hourly ambulatory systolic blood pressure and diastolic blood pressure readings
Change in Mean Ambulatory Blood Pressure from pre-intervention to 3-month follow-up | Change in Mean Ambulatory Blood Pressure assessed for 3 days at pre-intervention and three-month follow-up (an average of 18 weeks)
  Average of hourly ambulatory systolic blood pressure and diastolic blood pressure readings
Change in Momentary Positive Affect from pre-intervention to post-intervention | Change in Mean Momentary Positive Affect assessed for 3 days at pre-intervention and post-intervention (an average of 5 weeks)
  Average of state positive affect assessed hourly using 1-item scale, with scores ranging from 0-10 and higher scores indicating greater positive affect
Change in Momentary Positive Affect from pre-intervention to 3-month follow-up | Change in Mean Momentary Positive Affect assessed for 3 days at pre-intervention and three-month follow-up (an average of 18 weeks)
  Average of state positive affect assessed hourly using 1-item scale, with scores ranging from 0-10 and higher scores indicating greater positive affect
Change in Momentary Negative Affect from pre-intervention to post-intervention | Change in Mean Momentary Negative Affect assessed for 3 days at pre-intervention and post-intervention (an average of 5 weeks)
  Average of state negative affect assessed hourly using 1-item scale, with scores ranging from 0-10 and higher scores indicating greater negative affect
Change in Momentary Negative Affect from pre-intervention to 3-month follow-up | Change in Mean Momentary Negative Affect assessed for 3 days at pre-intervention and three-month follow-up (an average of 18 weeks)
  Average of state negative affect assessed hourly using 1-item scale, with scores ranging from 0-10 and higher scores indicating greater negative affect
Change in Negative Affect Reactivity to Task-Related Strain from pre-intervention to post-intervention | Change in Negative Affect Reactivity to Task Strain assessed for 3 days at pre-intervention and post-intervention (an average of 5 weeks)
  Average negative affect response (measured with 1-item scale) in relation to hourly measures of momentary strain (high task demand and low decision latitude)
Change in Negative Affect Reactivity to Task-Related Strain from pre-intervention to 3-month follow-up | Change in Negative Affect Reactivity to Task Strain assessed for 3 days at pre-intervention and three-month follow-up (an average of 18 weeks)
  Average negative affect response (measured with 1-item scale) in relation to hourly measures of momentary strain (high task demand and low decision latitude)
Change in Negative Affect Reactivity to Social Conflict from pre-intervention to post-intervention | Change in Negative Affect Reactivity to Social Conflict assessed for 3 days at pre-intervention and post-intervention (an average of 5 weeks)
  Average negative affect response (measured with 1-item scale) in relation to hourly measures of social conflict
Change in Negative Affect Reactivity to Social Conflict from pre-intervention to 3-month follow-up | Change in Negative Affect Reactivity to Social Conflict assessed for 3 days at pre-intervention and three-month follow-up (an average of 18 weeks)
  Average negative affect response (measured with 1-item scale) in relation to hourly measures of social conflict
Change in Blood Pressure Reactivity to Acute Stress from pre-intervention to post-intervention | Change in Blood Pressure Reactivity to Acute Stress from pre-intervention to post-intervention (average of 7 weeks)
  Assessed from blood pressure responses to an acute laboratory stress task
Change in Subjective Reactivity to Acute Stress from pre-intervention to post-intervention | Change in Subjective Reactivity to Acute Stress from pre-intervention to post-intervention (average of 7 weeks)
  Assessed via a 3-item measure of perceived stress to an acute laboratory stress task, with average score ranging from 0-100 and higher scores indicating greater stress
Change in Trait Affect from pre-intervention to post-intervention | Change in Trait Affect assessed at pre-intervention and post-intervention (average of 6 weeks)
  Assessed via the Trait Affect Scale (Cohen et al., 2003), a 25-item self-report questionnaire yielding three 3-item positive affect scales, three 3-item negative affect scales, one 4-item fatigue scale, and one 3-item fear scale, with average scores ranging from 0-4 and higher scores indicating greater positive affect, negative affect, fatigue, or fear
Change in Trait Affect from pre-intervention to 3-month follow-up | Change in Trait Affect assessed at pre-intervention and 3-month follow-up (average of 19 weeks)
  Assessed via the Trait Affect Scale (Cohen et al., 2003), a 25-item self-report questionnaire yielding three 3-item positive affect scales, three 3-item negative affect scales, one 4-item fatigue scale, and one 3-item fear scale, with average scores ranging from 0-4 and higher scores indicating greater positive affect, negative affect, fatigue, or fear
Change in Positive and Negative Social Exchanges from pre-intervention to post-intervention | Change in Social Exchanges from pre-intervention to post-intervention (average of 6 weeks)
  Assessed via that Positive and Negative Social Exchanges (PANSE), a 24-item measure that measures quality of interpersonal interactions, with two overall sum scores: Positive Social Exchanges, ranging from 0-48, with higher scores indicating more positive social exchanges, and Negative Social Exchanges, ranging from 0-48, with higher scores indicating more negative social exchanges; within each domain are 4 3-item subscales: informational support, instrumental support, companionship, emotional support, unwanted advice or intrusion, failure to provide help, unsympathetic or insensitive behavior, and rejection or neglect
Change in Positive and Negative Social Exchanges from pre-intervention to 3-month follow-up | Change in Social Exchanges from pre-intervention to 3-month follow-up (average of 19 weeks)
  Assessed via that Positive and Negative Social Exchanges (PANSE), a 24-item measure that measures quality of interpersonal interactions, with two overall sum scores: Positive Social Exchanges, ranging from 0-48, with higher scores indicating more positive social exchanges, and Negative Social Exchanges, ranging from 0-48, with higher scores indicating more negative social exchanges; within each domain are 4 3-item subscales: informational support, instrumental support, companionship, emotional support, unwanted advice or intrusion, failure to provide help, unsympathetic or insensitive behavior, and rejection or neglect
Change in Perceived Stress from pre-intervention to post-intervention | Change in Perceived Stress from pre-screening to post-intervention (average of 7 weeks)
  Assessed via the Perceived Stress Scale (PSS), a 10-item questionnaire that measures perceived stress over the past month, with total scores ranging from 0-40 and higher scores indicating greater perceived stress
Change in Perceived Stress from pre-intervention to 3-month follow-up | Change in Perceived Stress from pre-screening to three-month follow up (average of 20 weeks)
  Assessed via the Perceived Stress Scale (PSS), a 10-item questionnaire that measures perceived stress over the past month, with total scores ranging from 0-40 and higher scores indicating greater perceived stress
Change in Anxiety Symptoms from pre-intervention to post-intervention | Change in Anxiety Symptoms from pre-intervention to post-intervention (average of 6 weeks)
  Assessed via the Generalized Anxiety Disorder-7 (GAD-7), a 7-item measure of anxiety symptoms, with total score ranging from 0-21 and higher scores indicating greater anxiety severity
Change in Anxiety Symptoms from pre-intervention to 3-month follow-up | Change in Anxiety Symptoms from pre-intervention to three-month follow up (average of 19 weeks)
  Assessed via the Generalized Anxiety Disorder-7 (GAD-7), a 7-item measure of anxiety symptoms, with total score ranging from 0-21 and higher scores indicating greater anxiety severity
Change in Job Strain from pre-intervention to post-intervention | Change in Job Strain from pre-intervention to post-intervention (average of 6 weeks)
  Assessed via the Job Content Questionnaire (Karasek et al., 1985), a 42-item self-report instrument for employed individuals that measures (1) Work Demands (from 5 items measuring work load and intensity, with higher average scores indicating greater work demands) and (2) Decision Latitude (from a weighted sum of two subscales: Skill Discretion (6 items, with higher scores indicating greater creative challenge on the job) and Decision Authority (3 items, with higher scores indicating greater authority over day-to-day tasks)
Change in Job Strain from pre-intervention to 3-month follow-up | Change in Job Strain from pre-intervention to three-month follow up (average of 19 weeks)
  Assessed via the Job Content Questionnaire (Karasek et al., 1985), a 42-item self-report instrument for employed individuals that measures (1) Work Demands (from 5 items measuring work load and intensity, with higher average scores indicating greater work demands) and (2) Decision Latitude (from a weighted sum of two subscales: Skill Discretion (6 items, with higher scores indicating greater creative challenge on the job) and Decision Authority (3 items, with higher scores indicating greater authority over day-to-day tasks)
Daily Perceived Stress during mindfulness intervention | Collected daily throughout the 4-week intervention period for Mindfulness participants only
  Daily perceived stress (2-items from the Perceived Stress Scale) assessed daily via end-of-day diary during the mindfulness intervention period in the mindfulness condition only, with scores ranging from 0-10 and higher average scores indicating higher perceived stress, used to evaluate random vs. pre-selected prompt timing
Change in Momentary Perceived Stress before and after mindfulness prompts | Collected before and after mindfulness prompts throughout the 4-week intervention period for Mindfulness participants only
  Momentary perceived stress assessed via 1-item scale before and after each mindfulness prompt (delivered three times daily during the mindfulness intervention period in the mindfulness condition only), with scores ranging from 0-10 and higher average scores indicating higher perceived stress and greater change scores indicating greater reduction in perceived stress following mindfulness prompts
Mindfulness Prompt Helpfulness | Collected daily throughout the 4-week intervention period for Mindfulness participants only
  Helpfulness of daily mindfulness practice prompts assessed with 1-item in the mindfulness condition only, ranging from 0-10 with higher scores indicating greater helpfulness, used to evaluate random vs. pre-selected prompt timing

OTHER OUTCOMES:
Change in Momentary Perceived Stress | Change in Momentary Perceived Stress is assessed for 3 days at three timepoints: pre-intervention, post-intervention (an average of 5 weeks), and three-month follow-up (an average of 18 weeks)
  Average of state perceived stress assessed hourly using 2-items adapted from the Perceived Stress Scale, with scores ranging from 0-10 and higher scores indicating greater stress, and 1-item on current ongoing stress, with scores ranging from 0-10 and higher scores indicating greater stress
Change in Momentary Distress Tolerance | Change in Distress Tolerance assessed for 3 days at three timepoints: pre-intervention, post-intervention (an average of 5 weeks), and three-month follow-up (an average of 18 weeks)
  Average of state distress tolerance assessed hourly using 1-item scale with scores ranging from 0-10 and higher scores indicating greater distress intolerance
Change in Momentary Rumination | Change in Momentary Rumination is assessed for 3 days at three timepoints: pre-intervention, post-intervention (an average of 5 weeks), and three-month follow-up (an average of 18 weeks)
  Average of state rumination assessed hourly using 1-item scale with scores ranging from 0-10 and higher scores indicating greater rumination
Change in Daily Perceived Stress | Change in Daily Perceived Stress assessed for 7 days at three timepoints: pre-intervention, post-intervention (an average of 5 weeks), and three-month follow-up (an average of 18 weeks)
  Daily perceived stress (2-items from the Perceived Stress Scale) assessed daily via end-of-day diary, with average scores ranging from 0-10 and higher scores indicating greater stress
Change in Daily Positive Affect | Change in Mean Daily Positive Affect assessed for 7 days at three timepoints: pre-intervention, post-intervention (an average of 5 weeks), and three-month follow-up (an average of 18 weeks)
  Daily positive affect (composite of 3 positive affect items (calm, energetic, happy)) assessed daily via end-of-day diary, with average scores ranging from 0-10 and higher scores indicating greater positive affect
Change in Daily Negative Affect | Change in Mean Daily Negative Affect assessed for 7 days at three timepoints: pre-intervention, post-intervention (an average of 5 weeks), and three-month follow-up (an average of 18 weeks)
  Daily negative affect (composite of 3 negative affect items (angry, depressed, tense)) assessed daily via end-of-day diary, with average scores ranging from 0-10 and higher scores indicating greater negative affect
Change in Social Interactions | Change in frequency of Social Interactions assessed for 3 days at three timepoints: pre-intervention, post-intervention (an average of 5 weeks), and three-month follow-up (an average of 18 weeks)
  Frequency of social interactions assessed hourly using 1-item assessing current involvement in social interactions, 1-item assessing timing of most recent social interaction, and 1-item assessing number of social interactions
Change in Social Interaction Characteristics | Change in Social Interaction Characteristics assessed for 3 days at three timepoints: pre-intervention, post-intervention (an average of 5 weeks), and three-month follow-up (an average of 18 weeks)
  Characteristics of most recent social interaction assessed hourly using 4-item scale
Change in Social Interaction Responsiveness | Change in Social Interaction Responsiveness assessed for 3 days at three timepoints: pre-intervention, post-intervention (an average of 5 weeks), and three-month follow-up (an average of 18 weeks)
  Responsiveness of most recent social interaction assessed hourly using 2-item scale, with average scores ranging from 0-10 and higher scores indicating greater social interaction responsiveness
Change in Daily Loneliness | Change in Loneliness assessed for 7 days at three timepoints: pre-intervention, post-intervention (an average of 5 weeks), and three-month follow-up (an average of 18 weeks)
  Loneliness assessed daily using 1-item via end-of-day diary, with scores ranging from 0-10 and higher scores indicating greater loneliness
Change in Sleepiness | Change in Sleepiness assessed for 7 days at three timepoints: pre-intervention, post-intervention (an average of 5 weeks), and three-month follow-up (an average of 18 weeks)
  Sleepiness assessed daily using 2-items via end-of-day diary, with average scores ranging from 0-10 and higher scores indicating greater sleepiness
Change in Daily Life Mindfulness | Change in Daily Life Mindfulness assessed for 7 days at three timepoints: pre-intervention, post-intervention (an average of 5 weeks), and three-month follow-up (an average of 18 weeks)
  Mindful awareness assessed via end-of-day diary using 3-item scale, with average scores ranging from 0-10 and higher scores indicating greater mindfulness
Change in Daily Distress Tolerance | Change in Daily Distress Tolerance assessed for 7 days at three timepoints: pre-intervention, post-intervention (an average of 5 weeks), and three-month follow-up (an average of 18 weeks)
  Distress tolerance assessed via end-of-day diary using 1-item, with scores ranging from 0-10 and higher scores indicating greater distress tolerance
Change in Stressful Events | Change in Stressful Events assessed for 7 days at three timepoints: pre-intervention, post-intervention (an average of 5 weeks), and three-month follow-up (an average of 18 weeks)
  Stressful events assessed daily via end-of-day diary using 17-item scale
Change in Positive Events | Change in Positive Events assessed for 7 days at three timepoints: pre-intervention, post-intervention (an average of 5 weeks), and three-month follow-up (an average of 18 weeks)
  Positive events assessed daily via end-of-day diary using 7-item scale
Passive sensor stress models | Sensor data collected continuously for 7 days at three timepoints: pre-intervention, post-intervention (an average of 5 weeks), and three-month follow-up (an average of 18 weeks)
  Passive sensor data from smartphones (location, activity, screen status, battery, weather, time zone, communication) and wearable devices (heart rate, activity, sleep) combined to develop machine learning models predicting state stress
Change in Physical Activity | Change in Physical Activity assessed for 7 days at three timepoints: pre-intervention, post-intervention (an average of 5 weeks), and three-month follow-up (an average of 18 weeks)
  Average physical activity assessed via Fitbit estimate of caloric expenditure
Change in Sleep Duration | Change in Sleep Duration assessed for 7 days at three timepoints: pre-intervention, post-intervention (an average of 5 weeks), and three-month follow-up (an average of 18 weeks)
  Average sleep duration assessed via Fitbit
Change in Daily Sleep Patterns | Change in Sleep Patterns assessed for 3 days at three timepoints: pre-intervention, post-intervention (an average of 5 weeks), and three-month follow-up (an average of 18 weeks)
  Sleep patterns assessed each morning via 10-item questionnaire measuring sleep time and quality
Change in Self-Compassion | Change in Self-Compassion from pre-intervention to post-intervention (average of 6 weeks) and three-month follow up (average of 19 weeks)
  Assessed via the Self-Compassion Scale Short Form, a 12-item scale, with average scores ranging from 1-5 and higher scores indicating greater self-compassion
Change in Trait Mindfulness | Change in Trait Mindfulness from pre-intervention to post-intervention (average of 6 weeks) and three-month follow up (average of 19 weeks)
  Assessed via the Five Facet Mindfulness Questionnaire-Short Form, a 15-item scale with observing, describing, acting with awareness, nonreactivity, and nonjudgment subscales, with higher scores indicating higher mindfulness
Change in Experiential Avoidance | Change in Experiential Avoidance from pre-intervention to post-intervention (average of 6 weeks) and three-month follow up (average of 19 weeks)
  Assessed via the Acceptance and Action Questionnaire (AAQ-2), a 7-item scale assessing psychological inflexibility and experiential avoidance, with higher scores indicating higher avoidance
Change in Health Behaviors | Change in Health Behaviors from pre-intervention to post-intervention (average of 6 weeks) and three-month follow up (average of 19 weeks)
  Assessed using a 16-item measure that assesses general health behaviors (e.g., caffeine, smoking, alcohol, physical activity, sedentary behavior, diet)
Childhood Trauma | Pre-intervention, to be used in exploratory moderator analyses
  Assessed via the Childhood Trauma Questionnaire, a 28-item scale with 5 subscales (physical, sexual, and emotional abuse, and physical and emotional neglect), with higher scores indicating greater trauma
Everyday Discrimination | Pre-intervention, to be used in exploratory moderator analyses
  Assessed via the Everyday Discrimination Scale, a 10-item measure of perceived discrimination, with higher scores indicating higher discrimination
Continued Mindfulness Practice | Mindfulness Practice assessed for 7 days at two timepoints: post-intervention and three-month follow up
  Mindfulness practice after the intervention period assessed using a 2-item measure of duration and quality (mindfulness condition only) during end-of-day diary
Monthly Stress Management | Stress Management practice assessed monthly at post-intervention, 1-month follow-up, 2-month follow-up, and 3-month follow-up
  Stress management practice in the past month assessed via 5-item survey that asks participants to report on the type, frequency, and quality of practice, plus 2 items assessing psychological treatment and formal stress management during the study period at 3-month follow-up only

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W Kamarck, PhD, Principal Investigator — University of Pittsburgh; Emily K Lindsay, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to document and archive the data sets collected as part of this project to be made available in the public domain and on-line. Following publication of the primary aims, specific analyses and reporting, consolidated data, along with data dictionaries and program-specific setup syntax files, will be made publicly available via an online portal (e.g., Inter-university Consortium for Political and Social Research [ICPSR] data repository).
Time Frame: Final research data from this study will be deposited into the ICPSR repository approximately 6 to 12 months after the acceptance of peer-reviewed reports of results bearing on the project's specific aims.
Access Criteria: ICPSR will make the final research data from this project available to the broader social science research community. The ICPSR has policies and procedures in place that will provide data access to qualified researchers.